CLINICAL TRIAL: NCT04132622
Title: Low Dose Euthyrox in Treatments of Paraquat Intoxication: a Randomized, Controlled, Multicenter Trial in China.
Brief Title: Low Dose Euthyrox in Treatments of Paraquat Intoxication.
Acronym: LDETPI
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: First People's Hospital of Hangzhou (Other); Zhejiang Provincial Hospital of TCM (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CYM2019
Record Dates: First submitted 2019-10-17; First posted 2019-10-21 (Actual); Last update posted 2019-10-22 (Actual); Status verified 2019-10

CONDITIONS: Paraquat Poisoning
Keywords: Euthyrox; Paraquat Intoxication
MeSH Terms: interventions — Thyroxine

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Experimental therapy group (Experimental): Besides Traditional therapy，patients in this group will also receive thyroid replacement therapy.
  Interventions: Drug: Levothyroxine Sodium; Drug: Traditional therapy
- Traditional therapy group (Sham Comparator): Patients in Standard therapy group will receive treatments according to guideline worldwide.
  Interventions: Drug: Traditional therapy

INTERVENTIONS:
Drug: Levothyroxine Sodium — Levothyroxine Sodium Tablets (50 ug, calculated by Levothyroxine Sodium ), produced by Merck KGaA, Darmstadt.
  Other Names: Euthyrox, H20140052
  Arms: Experimental therapy group
Drug: Traditional therapy — including steroids, vitamin C, hemodialysis and blood perfusion.
  Other Names: Standard treatment

SUMMARY:
Paraquat is a common human toxicant and accounts for 20 deaths per million persons in the world. Paraquat usually cause multiple organ dysfunction syndrome, including liver, kidney, lung and heart dysfunction. Besides, pituitary insufficiency also occurs on those patients with paraquat poisoning, which leads to multiple endocrine gland dysfunction, involving adrenal gland, thyroid and sex gland.

As a result, the investigators decide to initiate the clinical trial to find whether thyroid replacement therapy can furtherly reduce the mortality, and improve patients long-term prognosis.

DETAILED DESCRIPTION:
Paraquat is a common human toxicant and accounts for 20 deaths per million persons in the world. Its accidental or deliberate ingestion is associated with a high mortality rate ranging from 40% to 70%. Paraquat usually cause multiple organ dysfunction syndrome, including liver, kidney, lung and heart dysfunction. Besides, pituitary insufficiency also occurs on those patients with paraquat poisoning, which leads to multiple endocrine gland dysfunction, involving adrenal gland, thyroid and sex gland. Nowadays, steroids, as a hormone replacement therapy, is one of most important drugs for paraquat poisoning, and it has decreased patients' mortality greatly since using it. However, the clinicians have not paid enough attention to thyroid replacement therapy, as thyroid dysfunction is also the key pathophysiological course when paraquat poisoning occurs.

As a result, the investigators decide to initiate the clinical trial to find whether thyroid replacement therapy can furtherly reduce the mortality, and improve patients long-term prognosis.

ELIGIBILITY:
Inclusion Criteria:

* all the patients who are diagnosed by paraquat poisoning

Exclusion Criteria:

* patients who can not cooperate with the trial; patients who would not like to join in the trial.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2020-01-01 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of death weekly | a week
  Rate of death in a week.
Rate of death monthly | a month
  Rate of death in a month.
Rate of death yearly | a year
  Rate of death in a year.
Survival rate yearly | a year
  Survival rate in a year.

SECONDARY OUTCOMES:
Number of Participants with Kidney dysfunction | a week, a month, a year
  Number of Participants with Kidney dysfunction with paraquat poisoning

CONTACTS AND LOCATIONS:
Overall Officials: Yuemei Chen, doctor, Study Chair — Second Affiliated Hospital of Zhejiang University School of Medicine

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hwang KY, Lee EY, Hong SY. Paraquat intoxication in Korea. Arch Environ Health. 2002 Mar-Apr;57(2):162-6. doi: 10.1080/00039890209602931. PMID 12194161
- [Background] Seok SJ, Gil HW, Jeong DS, Yang JO, Lee EY, Hong SY. Paraquat intoxication in subjects who attempt suicide: why they chose paraquat. Korean J Intern Med. 2009 Sep;24(3):247-51. doi: 10.3904/kjim.2009.24.3.247. Epub 2009 Aug 26. PMID 19721862
- [Background] Bismuth C, Garnier R, Baud FJ, Muszynski J, Keyes C. Paraquat poisoning. An overview of the current status. Drug Saf. 1990 Jul-Aug;5(4):243-51. doi: 10.2165/00002018-199005040-00002. PMID 2198050
- [Background] Kim SJ, Gil HW, Yang JO, Lee EY, Hong SY. The clinical features of acute kidney injury in patients with acute paraquat intoxication. Nephrol Dial Transplant. 2009 Apr;24(4):1226-32. doi: 10.1093/ndt/gfn615. Epub 2008 Nov 5. PMID 18987262
- [Background] Dinis-Oliveira RJ, Duarte JA, Sanchez-Navarro A, Remiao F, Bastos ML, Carvalho F. Paraquat poisonings: mechanisms of lung toxicity, clinical features, and treatment. Crit Rev Toxicol. 2008;38(1):13-71. doi: 10.1080/10408440701669959. PMID 18161502